CLINICAL TRIAL: NCT00595426
Title: A Phase 2b, Double-Blind, Double-Dummy, Randomized, Parallel Group Study to Evaluate the Safety and Efficacy of Twice Daily Dosing and Once Daily Dosing of YM150 in Subjects Undergoing Primary Elective Knee Arthroplasty
Brief Title: A Study to Evaluate the Safety and Efficacy of YM150 in Patients With Knee Replacement Surgery
Acronym: PEARL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 150-CL-033
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2010-05

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee Arthroplasty; Factor Xa; VTE; Thrombosis; Anticoagulants
MeSH Terms: conditions — Thrombosis | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1. YM150 Dose X, twice daily (Experimental)
  Interventions: Drug: YM150
- 2. YM150 Dose Y, once daily (Experimental)
  Interventions: Drug: YM150
- 3. YM150 Dose Y, twice daily (Experimental)
  Interventions: Drug: YM150
- 4. YM150 Dose Z, once daily (Experimental)
  Interventions: Drug: YM150
- 5. Warfarin (Active Comparator): various doses
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: YM150 — Oral
  Arms: 1. YM150 Dose X, twice daily; 2. YM150 Dose Y, once daily; 3. YM150 Dose Y, twice daily; 4. YM150 Dose Z, once daily
Drug: Warfarin — Oral
  Arms: 5. Warfarin

SUMMARY:
To evaluate the safety and efficacy of twice daily dosing and once daily dosing of YM150 in subjects undergoing primary elective knee replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for elective primary knee arthroplasty
* Written Informed consent obtained

Exclusion Criteria:

* Subject has documented history of previous VTE
* Subject is considered to be at increased risk of VTE
* Subject has active bleeding or any condition associated with increased risk of bleeding
* Subject is planning to have surgery on the contralateral knee at the same time or within 6 weeks after enrollment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The incidence of total venous thromboembolisms (VTE). | 6 Weeks
The incidence of bleeding events classified as major by the Adjudication Committee | 6 Weeks

SECONDARY OUTCOMES:
Evaluation of efficacy variables including: Proximal VTE, Distal VTE, Confirmed symptomatic VTE, death due to any cause | 6 Weeks
Incidence of the bleeding types: major, clinically relevant nonmajor, minor | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (48):
- United States (38):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Fountain Valley, California
  - La Mesa, California
  - Long Beach, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Yuba City, California
  - Aurora, Colorado
  - Denver, Colorado
  - Lone Tree, Colorado
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Bradenton, Florida
  - Gulf Breeze, Florida
  - Hollywood, Florida
  - St. Petersburg, Florida
  - Decatur, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Springfield, Illinois
  - Baltimore, Maryland
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Canada (10):
  - Red Deer, Alberta
  - Ajax, Ontario
  - Burlington, Ontario
  - Montreal, Ontario
  - Newmarket, Ontario
  - Saint Catherines, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Waterloo, Ontario
  - Charlottetown, Prince Edward Island